CLINICAL TRIAL: NCT03780426
Title: Transcranial Static Magnetic Field Stimulation (tSMS) in Essential Tremor
Brief Title: tSMS in Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación de investigación HM (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Fundacion de Investigación HM
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tSMS left motor cortex (sham right) (Experimental): 30 min of tSMS applied to the left motor cortex with sham on the right motor cortex
  Interventions: Device: tSMS; Device: sham
- tSMS right motor cortex (sham left) (Experimental): 30 min of tSMS applied to the right motor cortex with sham on the left motor cortex
  Interventions: Device: tSMS; Device: sham

INTERVENTIONS:
Device: tSMS — Transcranial static magnetic field stimulation (tSMS) is a non-invasive brain stimulation (NIBS) technique that decreases cortical excitability (Oliviero et al., 2011; Oliviero et al., 2015; Dileone et al., 2018). Static magnetic fields suitable for tSMS are obtained with commercially available neodymium magnets. We will use a cylindrical neodymium magnet of 45 mm diameter and 30 mm of thickness, with a weight of 360 g (MAG45r; Neurek SL, Toledo, Spain), which will be applied with south polarity to the left or right motor cortex, using a tSMS helmet (MAGmv1.0; Neurek SL, Toledo, Spain).
  Other Names: MAGmv1.0 with MAG45r, Neurek S.L. (Toledo, Spain)
Device: sham — A non-magnetic metal cylinder, with the same size, weight and appearance of the magnet, will be used for sham stimulation (MAG45s; Neurek SL, Toledo, Spain) of motor cortex contralateral to the stimulated hemisphere.
  Other Names: MAGmv1.0 with MAG45s, Neurek S.L. (Toledo, Spain)

SUMMARY:
This is randomized double-blind study to study the hypothesis that transcranial static magnetic field stimulation of the primary motor cortex improves tremor in patients with essential tremor. Half of the patients will receive tSMS of the left hemisphere and the other half of the right hemisphere.

ELIGIBILITY:
Inclusion Criteria:

* Essential tremor

Exclusion Criteria:

* MRI-incompatible metal objects in the body (e.g. cardiac pacemakers)
* other main neuropsychiatric co-morbidity
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in postural tremor amplitude in the hand contralateral to hemispheren that received tSMS treatment compared to the hand contralateral to the hemisphere that received sham treatment, as measured by accelerometry. | Immediately after treatment compared baseline

SECONDARY OUTCOMES:
Change from baseline in postural tremor amplitude 15 minutes after treatment, as measured by accelerometry. | 15 minutes after treatment compared to baseline
Change from baseline in rest tremor amplitude, as measured by accelerometry. | Immediately after treatment and 15 minutes after treatment compared baseline.
Change from baseline in tremor frequency, as measured by accelerometry. | Immediately after treatment and 15 minutes after treatment compared baseline.
Change from baseline in the Clinical Rating Scale for Tremor part B (drawing) | 5 minutes after treatment and 20 minutes after treatment compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CINAC, Hospital Universitario Puerta del Sur, Móstoles, Madrid, Spain

REFERENCES:
- [Background] Oliviero A, Mordillo-Mateos L, Arias P, Panyavin I, Foffani G, Aguilar J. Transcranial static magnetic field stimulation of the human motor cortex. J Physiol. 2011 Oct 15;589(Pt 20):4949-58. doi: 10.1113/jphysiol.2011.211953. Epub 2011 Aug 1. PMID 21807616
- [Background] Oliviero A, Carrasco-Lopez MC, Campolo M, Perez-Borrego YA, Soto-Leon V, Gonzalez-Rosa JJ, Higuero AM, Strange BA, Abad-Rodriguez J, Foffani G. Safety Study of Transcranial Static Magnetic Field Stimulation (tSMS) of the Human Cortex. Brain Stimul. 2015 May-Jun;8(3):481-5. doi: 10.1016/j.brs.2014.12.002. Epub 2014 Dec 11. PMID 25595064
- [Background] Dileone M, Mordillo-Mateos L, Oliviero A, Foffani G. Long-lasting effects of transcranial static magnetic field stimulation on motor cortex excitability. Brain Stimul. 2018 Jul-Aug;11(4):676-688. doi: 10.1016/j.brs.2018.02.005. Epub 2018 Feb 7. PMID 29500043
- [Derived] Urso D, Monje MHG, Fernandez-Rodriguez B, Vela-Desojo L, Oliviero A, Foffani G, Ammann C. Transcranial static magnetic field stimulation of the primary motor cortex in essential tremor: a randomized pilot study. NPJ Parkinsons Dis. 2025 Nov 26;11(1):336. doi: 10.1038/s41531-025-01182-x. PMID 41298510